CLINICAL TRIAL: NCT01742507
Title: A Randomized Optical Coherence Tomography Study Comparing Resolute Integrity to Biomatrix Drug-eluting Stent on the Degree of Early Stent Healing and Late Lumen Loss.The OCT-ORION Study
Brief Title: A Study Comparing Two Stent on the Degree of Early Stent Healing and Late Lumen Loss.The OCT-ORION Study
Acronym: OCT-ORION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Stephen Lee, Professor and Chief of Cardiology, The University of Hong Kong
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 12-093
Record Dates: First submitted 2012-03-22; First posted 2012-12-05 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Coronary Artery Disease
Keywords: Stent, OCT
MeSH Terms: conditions — Coronary Artery Disease; Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medtronic Resolute Integrity Stent (Active Comparator): Medtronic Resolute Integrity Stent
  Interventions: Device: Resolute Integrity Stent
- Biomatrix stent (Active Comparator): Biomatrix stent
  Interventions: Device: Biomatrix stent

INTERVENTIONS:
Device: Resolute Integrity Stent — Resolute Integrity Stent
  Arms: Medtronic Resolute Integrity Stent
Device: Biomatrix stent — Biomatrix stent
  Arms: Biomatrix stent

SUMMARY:
Stent coverage and neo-intimal growth can be evaluated in-detail by intracoronary optical coherence tomography (OCT), which is a catheter-based imaging technique. It is performed as part of the PCI procedure. OCT is the optical analogue of intravascular ultrasound (IVUS), except that it can provide much higher resolution of coronary cross sectional images than IVUS. The LightLab C7XR OCT system (Frequency Domain OCT) used in this Hospital has obtained full CE Mark, approved by the US FDA, and approved for clinical use in Hong Kong. It has been shown to be safe in clinical settings and has been used in over 300 patients without complication at Queen Mary Hospital.

In this study, stent coverage and neo-intimal growth between zotarolimus-eluting stents (ZES) and biolimus-eluting stents (BES) will be compared by using OCT at 9 month and specific post-intervention re-study intervals.

The investigators objective is to investigate the clinical impact and OCT difference on early stent healing and late lumen loss between the two new-generation limus-eluting-stents - Resolute Integrity and Biomatrix, which differ in stent design, eluting drug and coating polymer.

DETAILED DESCRIPTION:
This is a prospective, randomised, assessor-blinded, single centre study. Patients with symptomatic coronary artery diseases in 2 or 3 coronary vessels requiring PCI are eligible for the study. PCI will be performed in the usual manner to all the study lesions in the same procedure. In a randomized fashion, each patient will have one artery with critical disease(s) treated by the Resolute Integrity Stent(s) and the other artery treated by the Biomatrix Stent(s).

Baseline OCT data will be obtained right after stenting. The remaining coronary artery, if diseased and required PCI treatment, will be treated during the angiographic and OCT follow-up as a staged procedure. Patients will be randomly assigned into 5 groups with equal number, receiving a follow-up coronary angiogram with OCT from 2, 3, 4, 5 and 6 months interval post-intervention. Each patient will serve as his/her own control comparing the 2 types of stents. At 9-month post-intervention, all patients will receive a second follow-up coronary angiogram with OCT. All OCT data analyses will be performed in a blinded fashion by a core laboratory. Phone follow up will be carried out for cardiac events at 1 year and 2 year of post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-85 years old
* Patient with symptomatic coronary artery diseases involving two or more vessels requiring percutaneous coronary intervention

Exclusion Criteria:

* Patient who is unable to give consent
* Patient in acute myocardial infarction or unstable angina
* Patient who is hemodynamically unstable
* Patient who is allergic to contrast agents
* Patient who is allergic to anti-platelet agents
* Patient who is allergic to zotarolimus
* Patient who is allergic to biolimus
* Patient who is pregnant
* Patient who has planned surgery in the following 12 months after percutaneous coronary intervention
* Left main coronary lesion
* Bifurcation lesion
* Chronic total occlusion lesion
* Coronary vessel size smaller than 2.5mm
* Coronary lesion longer than 38mm in length

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
• OCT derived percentage stent strut coverage at 9 month | 9 month
  OCT derived percentage stent strut coverage at 9 month

SECONDARY OUTCOMES:
Angiographic binary stenosis | 9 month
  • Angiographic binary stenosis at 9 month
• OCT derived neo-intimal area at 9 month | at 9 month
  • OCT derived neo-intimal area at 9 month
• Minimal lumen diameter by Quantitative Coronary Analysis (QCA) at 9 month | 9 month
  • Minimal lumen diameter by Quantitative Coronary Analysis (QCA) at 9 month
• All major adverse cardiac events (all cardiac deaths, myocardial infarction, target vessel failure and target lesion revascularization, and stent thrombosis) at the pre-defined 2 to 9 months angiographic and OCT follow-up. | 2 to 9 months
  • All major adverse cardiac events (all cardiac deaths, myocardial infarction, target vessel failure and target lesion revascularization, and stent thrombosis) at the pre-defined 2 to 9 months angiographic and OCT follow-up.
• Target vessel stent thrombosis per Academic Research Consortium (ARC) definition | from enrollment till 2 years follow up
  • Target vessel stent thrombosis per Academic Research Consortium (ARC) definition
Percentage of stent strut malapposition | 9 month
  Percentage of stent strut malapposition
Mean neo-intimal thickness (NIT) at 9 month | 9 month
  Mean neo-intimal thickness (NIT) at 9 month
Stent volume | at 9 month
  Stent volume
Lumen volume | at 9 month
  Lumen volume
Neointimal Hyperplasia (NIH) volume | at 9 month
  Neointimal Hyperplasia (NIH) volume

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wai Luen LEE, MD FRCP FACC, Principal Investigator — Queen Mary Hosptial, The Univeristy of Hong Kong
Locations (1):
- Division of Cardiology, Department of Medicine, QMH, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Result] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Result] Stone GW, Ellis SG, Cox DA, Hermiller J, O'Shaughnessy C, Mann JT, Turco M, Caputo R, Bergin P, Greenberg J, Popma JJ, Russell ME; TAXUS-IV Investigators. A polymer-based, paclitaxel-eluting stent in patients with coronary artery disease. N Engl J Med. 2004 Jan 15;350(3):221-31. doi: 10.1056/NEJMoa032441. PMID 14724301
- [Result] Kastrati A, Mehilli J, Pache J, Kaiser C, Valgimigli M, Kelbaek H, Menichelli M, Sabate M, Suttorp MJ, Baumgart D, Seyfarth M, Pfisterer ME, Schomig A. Analysis of 14 trials comparing sirolimus-eluting stents with bare-metal stents. N Engl J Med. 2007 Mar 8;356(10):1030-9. doi: 10.1056/NEJMoa067484. Epub 2007 Feb 12. PMID 17296823
- [Result] Stone GW, Moses JW, Ellis SG, Schofer J, Dawkins KD, Morice MC, Colombo A, Schampaert E, Grube E, Kirtane AJ, Cutlip DE, Fahy M, Pocock SJ, Mehran R, Leon MB. Safety and efficacy of sirolimus- and paclitaxel-eluting coronary stents. N Engl J Med. 2007 Mar 8;356(10):998-1008. doi: 10.1056/NEJMoa067193. Epub 2007 Feb 12. PMID 17296824
- [Result] Bavry AA, Kumbhani DJ, Helton TJ, Borek PP, Mood GR, Bhatt DL. Late thrombosis of drug-eluting stents: a meta-analysis of randomized clinical trials. Am J Med. 2006 Dec;119(12):1056-61. doi: 10.1016/j.amjmed.2006.01.023. PMID 17145250
- [Result] Matsumoto D, Shite J, Shinke T, Otake H, Tanino Y, Ogasawara D, Sawada T, Paredes OL, Hirata K, Yokoyama M. Neointimal coverage of sirolimus-eluting stents at 6-month follow-up: evaluated by optical coherence tomography. Eur Heart J. 2007 Apr;28(8):961-7. doi: 10.1093/eurheartj/ehl413. Epub 2006 Nov 29. PMID 17135281
- [Result] Kim JS, Fan C, Choi D, Jang IK, Lee JM, Kim TH, Park SM, Paik SI, Ko YG, Hong MK, Jang Y, Chung N. Different patterns of neointimal coverage between acute coronary syndrome and stable angina after various types of drug-eluting stents implantation; 9-month follow-up optical coherence tomography study. Int J Cardiol. 2011 Feb 3;146(3):341-6. doi: 10.1016/j.ijcard.2009.07.012. Epub 2009 Aug 25. PMID 19709765
- [Result] Barlis P, Regar E, Serruys PW, Dimopoulos K, van der Giessen WJ, van Geuns RJ, Ferrante G, Wandel S, Windecker S, van Es GA, Eerdmans P, Juni P, di Mario C. An optical coherence tomography study of a biodegradable vs. durable polymer-coated limus-eluting stent: a LEADERS trial sub-study. Eur Heart J. 2010 Jan;31(2):165-76. doi: 10.1093/eurheartj/ehp480. Epub 2009 Nov 4. PMID 19889649
- [Result] Udipi K, Melder RJ, Chen M, Cheng P, Hezi-Yamit A, Sullivan C, Wong J, Wilcox J. The next generation Endeavor Resolute Stent: role of the BioLinx Polymer System. EuroIntervention. 2007 May;3(1):137-9. No abstract available. PMID 19737697
- [Result] Serruys PW, Silber S, Garg S, van Geuns RJ, Richardt G, Buszman PE, Kelbaek H, van Boven AJ, Hofma SH, Linke A, Klauss V, Wijns W, Macaya C, Garot P, DiMario C, Manoharan G, Kornowski R, Ischinger T, Bartorelli A, Ronden J, Bressers M, Gobbens P, Negoita M, van Leeuwen F, Windecker S. Comparison of zotarolimus-eluting and everolimus-eluting coronary stents. N Engl J Med. 2010 Jul 8;363(2):136-46. doi: 10.1056/NEJMoa1004130. Epub 2010 Jun 16. PMID 20554978
- [Result] Silber S, Windecker S, Vranckx P, Serruys PW; RESOLUTE All Comers investigators. Unrestricted randomised use of two new generation drug-eluting coronary stents: 2-year patient-related versus stent-related outcomes from the RESOLUTE All Comers trial. Lancet. 2011 Apr 9;377(9773):1241-7. doi: 10.1016/S0140-6736(11)60395-4. Epub 2011 Apr 1. PMID 21459430
- [Result] Grube E, Buellesfeld L. BioMatrix Biolimus A9-eluting coronary stent: a next-generation drug-eluting stent for coronary artery disease. Expert Rev Med Devices. 2006 Nov;3(6):731-41. doi: 10.1586/17434440.3.6.731. PMID 17280537
- [Result] Grube E, Hauptmann KE, Buellesfeld L, Lim V, Abizaid A. Six-month results of a randomized study to evaluate safety and efficacy of a Biolimus A9 eluting stent with a biodegradable polymer coating. EuroIntervention. 2005 May;1(1):53-7. PMID 19758877
- [Result] Windecker S, Serruys PW, Wandel S, Buszman P, Trznadel S, Linke A, Lenk K, Ischinger T, Klauss V, Eberli F, Corti R, Wijns W, Morice MC, di Mario C, Davies S, van Geuns RJ, Eerdmans P, van Es GA, Meier B, Juni P. Biolimus-eluting stent with biodegradable polymer versus sirolimus-eluting stent with durable polymer for coronary revascularisation (LEADERS): a randomised non-inferiority trial. Lancet. 2008 Sep 27;372(9644):1163-73. doi: 10.1016/S0140-6736(08)61244-1. Epub 2008 Aug 31. PMID 18765162
- [Result] Yamaguchi T, Terashima M, Akasaka T, Hayashi T, Mizuno K, Muramatsu T, Nakamura M, Nakamura S, Saito S, Takano M, Takayama T, Yoshikawa J, Suzuki T. Safety and feasibility of an intravascular optical coherence tomography image wire system in the clinical setting. Am J Cardiol. 2008 Mar 1;101(5):562-7. doi: 10.1016/j.amjcard.2007.09.116. Epub 2008 Jan 10. PMID 18307999
- [Result] Prati F, Cera M, Ramazzotti V, Imola F, Giudice R, Albertucci M. Safety and feasibility of a new non-occlusive technique for facilitated intracoronary optical coherence tomography (OCT) acquisition in various clinical and anatomical scenarios. EuroIntervention. 2007 Nov;3(3):365-70. doi: 10.4244/eijv3i3a66. PMID 19737719
- [Derived] Lee SWL, Tam FCC, Lam SCC, Kong SL, Shea CP, Chan KKW, Wong MKL, Chan MPH, Wong AYT, Yung ASY, Lam YM, Zhang LW, Wu KKY, Mintz GS, Maehara A. The OCT-ORION Study: A Randomized Optical Coherence Tomography Study Comparing Resolute Integrity to Biomatrix Drug-Eluting Stent on the Degree of Early Stent Healing and Late Lumen Loss. Circ Cardiovasc Interv. 2018 Apr;11(4):e006034. doi: 10.1161/CIRCINTERVENTIONS.117.006034. PMID 29654119